CLINICAL TRIAL: NCT02228096
Title: A Phase II, Single Arm, Multicenter Trial to Determine the Efficacy and Safety of CTL019 in Pediatric Patients With Relapsed and Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: Study of Efficacy and Safety of CTL019 in Pediatric ALL Patients
Acronym: ENSIGN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019B2205J; 2015-003736-13 (EudraCT Number)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Relapsed B-cell Acute Lymphoblastic Leukemia; Refractory B-cell Acute Lymphoblastic Leukemia
Keywords: relapsed/refractory; Philadelphia chromosome positive acute lymphoblastic leukemia; Pharmaceuticals; Philadelphia chromosome positive; Acute Lymphoid Leukemia (ALL); Acute Lymphocytic Leukemia (ALL); CTL019; tisagenlecleucel
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tisagenlecleucel (CTL019) (Experimental): Pediatric patients with relapsed/refractory B-cell ALL
  Interventions: Biological: CTL019 T-cells

INTERVENTIONS:
Biological: CTL019 T-cells — A target dose of CTL019 transduced cells will consist of a single infusion of 2.0 to 5.0 x 10^6 CTL019 transduced cells per kg body weight (for patients ≤ 50 kg) and 1.0 to 2.5 x 10^8 CTL019 transduced viable T cells (for patients > 50 kg). The following cell dose ranges may be infused if all other safety release criteria are met: 0.2 to 5.0 x 10^6 CTL019 transduced viable T cells per kg body weight (for patient ≤ 50 kg) and 0.1 to 2.5 x 10^8 CTL019 transduced viable T cells (for patients > 50 kg).
  Other Names: tisagenlecleucel

SUMMARY:
This was a single arm, open-label, multi-center, phase II study to determine the efficacy and safety of an experimental therapy called CTL019 T-cells in pediatric patients with B-cell acute lymphoblastic leukemia, who were refractory to standard chemotherapy regimen or relapsed after allogeneic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory pediatric B-cell ALL and lymphoblastic lymphoma:

  1. 2nd or greater Bone Marrow (BM) relapse OR
  2. Any BM relapse after allogeneic SCT and must be > 6 months from SCT at the time of CTL019 infusion OR
  3. Refractory as defined by not achieving a CR after 2 cycles of a standard chemotherapy regimen chemotherapy regimen or chemorefractory as defined by not achieving a CR after 1 cycle of standard chemotherapy for relapse leukemia OR
  4. Patients with Philadelphia chromosome positive (Ph+) ALL are eligible if they are intolerant to or have failed 2 lines of tyrosine kinase inhibitor therapy (TKI), or if TKI therapy is contraindicated OR
  5. Ineligible for allogeneic SCT
* For relapsed patients, CD19 tumor expression demonstrated in bone marrow or peripheral blood by flow cytometry within 3 months of study entry
* Adequate organ function defined as:

  1. Renal function defined as (Calculated creatinine clearance or radioisotope Glomerular Filtration Rate (GFR) > 60 mL/min/1.73 m2 OR serum creatinine based on age/gender
  2. Alanine Aminotransferase (ALT) <= 5 times the upper limit of normal (ULN) for age;
  3. Bilirubin < 2.0 mg/dL;
  4. Must have a minimum level of pulmonary reserve defined as ≤Grade 1 dyspnea and pulse oxygenation > 91% on room air
  5. Left Ventricular Shortening Fraction (LVSF) ≥ 28% confirmed by echocardiogram, or Left Ventricular Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram or MUGA within 7 days of screening
* Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening
* Life expectancy > 12 weeks
* Age 3 at the time of screening per protocol to age 21 at the time of initial diagnosis
* Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) performance status ≥ 50 at screening
* Signed written informed consent and assent forms (if applicable) must be obtained prior to any study procedures
* Once all other eligibility criteria are confirmed, must have an apheresis product of non-mobilized cells received and accepted by the manufacturing site. Note: Apheresis product will not be shipped to or assessed for acceptance by the manufacturing site until documented confirmation of all other eligibility criteria is received.
* Patients with active CNS leukemia involvement defined as CNS-3 by CSF findings only are eligible but will have their CTL019 infusion delayed until CNS disease is reduced to CNS-1 or CNS-2 by CSF findings. Patients with other forms of active CNS-3 leukemic involvement such as CNS parenchymal or ocular disease, cranial nerve involvement or significant leptomeningeal disease are not eligible. However, such patients with other forms of CNS-3 leukemic involvement (non-CSF involvement) are eligible if there is documented evidence of disease stabilization for at least 3 months prior to CTL019 infusion. Patients must have no acute/ongoing neurologic toxicity > Grade 1 with the exception of a history of controlled seizures or fixed neurologic deficits that have been stable/improving over the past 3 months.

Exclusion Criteria:

* Isolated extra-medullary disease relapse
* Patients with concomitant genetic syndrome: such as patients with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Patients with Down Syndrome will not be excluded.
* Patients with Burkitt's lymphoma/leukemia (i.e. patients with mature B-cell ALL, leukemia with B-cell [surface Immunoglobulin (sIg) positive and kappa or lambda restricted positivity] ALL, with FAB L3 morphology and /or a MYC translocation)
* Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
* Prior treatment with gene therapy product
* Treatment with any prior anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD)
* Patient has participated in an investigational research study using an investigational agent within the last 30 days prior to screening
* Pregnant or nursing (lactating) women. NOTE: female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
* Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening
* HIV positive test within 8 weeks of screening
* The following medications are excluded:

  1. Steroids: Therapeutic systemic doses of steroids must be stopped > 72 hours prior to CTL019 infusion. However, the following physiological replacement doses of steroids are allowed: < 12 mg/m2/day hydrocortisone or equivalent
  2. Allogeneic cellular therapy: Any donor lymphocyte infusions (DLI) must be completed > 6 weeks prior to CTL019 infusion
  3. GVHD therapies: Any systemic drug used for GVHD must be stopped > 4 weeks prior to CTL019 infusion to confirm that GVHD recurrence is not observed (e.g. calcineurin inhibitors, methotrexate or other chemotherapy drugs, mycophenolate, rapamycin, thalidomide, or immunosuppressive antibodies such as anti-CD20 (rituximab), anti-tumor necrosis factor [anti-TNF], anti-interleukin 6 [anti-IL6] or anti-interleukin 6 receptor [anti-IL6R], systemic steroids)
  4. Chemotherapy:
* Tyrosine kinase inhibitors and hydroxyurea must be stopped > 72 hours prior to CTL019 infusion
* The following drugs must be stopped > 1 week prior to CTL019 infusion and should not be administered concomitantly or following lymphodepleting chemotherapy: vincristine, 6-mercaptopurine, 6-thioguanine, methotrexate < 25 mg/m2, cytosine arabinoside < 100 mg/m2/day, asparaginase (non-pegylated)
* The following drugs must be stopped >2 weeks prior to CTL019 infusion: salvage chemotherapy (e.g. clofarabine, cytosine arabinoside > 100 mg/m2, anthracyclines, cyclophosphamide, methotrexate ≥ 25 mg/m2), excluding the required lymphodepleting chemotherapy drugs
* Pegylated-asparaginase must be stopped > 4 weeks prior to CTL019 infusion e. CNS disease prophylaxis:
* CNS prophylaxis treatment must be stopped > 1 week prior to CTL019 infusion (e.g. intrathecal methotrexate) f. Radiotherapy:
* Non-CNS site of radiation must be completed > 2 weeks prior to CTL019 infusion
* CNS directed radiation must be completed > 8 weeks prior to CTL019 infusion g. Anti T-cell Antibodies: Administration of any T cell lytic or toxic antibody (e.g. alemtuzumab) within 8 weeks prior to CTL019 is prohibited since residual lytic levels may destroy the infused CTL019 cells and/or prevent their in vivo expansion. If such an agent has been administered within 8 weeks prior to CTL019, contact the Sponsor, consider consultation with an pharmacology expert, and consider measuring residual drug levels, if feasible, prior to CTL019 infusion Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) and all male participants, unless they are using highly effective methods of contraception for a period of 1 year after the CTL019 infusion. Highly effective contraception methods include:

  1. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are NOT acceptable methods of contraception
  2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  3. Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient
  4. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
  5. Use of IUDs are excluded due to increased risks of infection and bleeding in this population. However, IUD inserted prior to consent may remain in place, and a second method of contraception is mandated
  6. In case of use of oral contraception, women must be stable on the same pill for a minimum of 3 months before taking study treatment.

Women who are not of reproductive potential (defined as either <11 years of age, Tanner Stage 1, post-menopausal for at least 24 consecutive months (i.e. have had no menses) or have undergone hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy) are eligible without requiring the use of contraception. Women who are not yet of reproductive potential are to agree to use acceptable forms of contraception when they reach reproductive potential if within 1 year of CTL019 or if CAR cells are present in the blood by PCR. Acceptable documentation includes written or oral documentation communicated by clinician or clinician's staff of one of the following:

1. Demographics show age < 11
2. Physical examination indicates Tanner Stage 1
3. Physician report/letter
4. Operative report or other source documentation in the patient record
5. Discharge summary
6. Follicle stimulating hormone measurement elevated into the menopausal range

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (13):
  - Childrens Hospital Los Angeles SC, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Children's Healthcare of Atlanta SC-2, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mercy Children's Kansas University, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oregon Health and Science University SC, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center SC, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Laetsch TW, Maude SL, Balduzzi A, Rives S, Bittencourt H, Boyer MW, Buechner J, De Moerloose B, Qayed M, Phillips CL, Pulsipher MA, Hiramatsu H, Tiwari R, Grupp SA. Tisagenlecleucel in pediatric and young adult patients with Down syndrome-associated relapsed/refractory acute lymphoblastic leukemia. Leukemia. 2022 Jun;36(6):1508-1515. doi: 10.1038/s41375-022-01550-z. Epub 2022 Apr 14. PMID 35422096
- [Derived] Thudium Mueller K, Grupp SA, Maude SL, Levine JE, Pulsipher MA, Boyer MW, August KJ, Myers GD, Tam CS, Jaeger U, Foley SR, Borchmann P, Schuster SJ, Waller EK, Awasthi R, Potthoff B, Warren A, Waldron ER, McBlane F, Chassot-Agostinho A, Laetsch TW. Tisagenlecleucel immunogenicity in relapsed/refractory acute lymphoblastic leukemia and diffuse large B-cell lymphoma. Blood Adv. 2021 Dec 14;5(23):4980-4991. doi: 10.1182/bloodadvances.2020003844. PMID 34432863
- [Derived] Levine JE, Grupp SA, Pulsipher MA, Dietz AC, Rives S, Myers GD, August KJ, Verneris MR, Buechner J, Laetsch TW, Bittencourt H, Baruchel A, Boyer MW, De Moerloose B, Qayed M, Davies SM, Phillips CL, Driscoll TA, Bader P, Schlis K, Wood PA, Mody R, Yi L, Leung M, Eldjerou LK, June CH, Maude SL. Pooled safety analysis of tisagenlecleucel in children and young adults with B cell acute lymphoblastic leukemia. J Immunother Cancer. 2021 Aug;9(8):e002287. doi: 10.1136/jitc-2020-002287. PMID 34353848
- [Derived] Buechner J, Grupp SA, Hiramatsu H, Teachey DT, Rives S, Laetsch TW, Yanik GA, Wood P, Awasthi R, Yi L, Chassot-Agostinho A, Eldjerou LK, De Moerloose B. Practical guidelines for monitoring and management of coagulopathy following tisagenlecleucel CAR T-cell therapy. Blood Adv. 2021 Jan 26;5(2):593-601. doi: 10.1182/bloodadvances.2020002757. PMID 33496754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 14-Aug-2014 (FPFV) and 22-Sep-2017 (LPFV). At the time of LPLV (24-May-2019), the sponsor had decided to transfer all ongoing patients to a separate long-term follow-up study to complete the planned 15 years of follow-up. These patients are designated with the reason for discontinuation as "terminated by sponsor".
Pre-assignment Details: "Enrolled" means all eligibility criteria were met and apheresis was accepted by the manufacturing facility. Patients could discontinue the trial after enrollment and prior to tisagenlecleucel infusion. Although 75 patients were enrolled, only 64 were infused as 11 discontinued prior to infusion.
Groups:
- Tisagenlecleucel (CTL019) - All Participants: Pediatric participants with r/r B-cell who were infused with tisagenlecleucel
Period: Overall Study
Arm/Group | Tisagenlecleucel (CTL019) - All Participants
Started | 75
Enrolled Into Long-term f/u Protocol | 31
Enrolled But Not Infused (Enrolled means all eligibility criteria were met & apheresis was accepted by manufacturing facility) | 11
Enrolled and Infused | 64
Completed | 4 (Completed = study follow-up completed)
Not Completed | 71
Not completed — Study terminated by Sponsor | 24
Not completed — Lack of Efficacy | 18
Not completed — Death | 12
Not completed — Physician Decision | 3
Not completed — Subject/guardian decision | 2
Not completed — New therapy for study indication | 1
Not completed — Enrolled, not infused | 11

BASELINE CHARACTERISTICS:
Population: Enrolled Set: All participants who met all the inclusion/exclusion criteria, and whose apheresis product is received and accepted by the manufacturing facilty
Groups:
- Not Infused: Pediatric patients with r/r B-cell who were enrolled in the study but not infused with tisagenlecleucel
- Total: Total of all reporting groups
Arm/Group | Tisagenlecleucel (CTL019) - All Participants | Not Infused | Total
Number analyzed (Participants) | 64 | 11 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.4 (5.16) | 15.2 (5.44) | 12.8 (5.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 1 | 35
  Male | 30 | 10 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  White | 52 | 8 | 60
  Asian | 5 | 1 | 6
  Other | 7 | 2 | 9
Weight [Mean (Standard Deviation); unit: kg] | 43.7 (20.10) | 86.2 (41.52) | 47.3 (25.25)
Karnofsky/Lansky performance status [Count of Participants; unit: Participants] — Karnofsky/Lansky performance status helps determine the functional status of a recipient. This status is a critical data field that has been determined to be essential for all outcome-based analyses. Karnofsky Scale: designed for recipients aged 16 years & older; Lansky Scale: designed for recipients 1 year old to less than 16 years old. The Karnofsky/Lansky performances are based from 100 to 0, where 100 is "perfect" health & 0 is death. The scale: Able to carry on normal activity, no special care needed (80- 100); Mild to moderate restriction (50-70); Moderate to severe restriction (10- 40). Population: FAS = All subjects who received an infusion of tisagenlecleucel
  Participants
    100: number analyzed (Participants) | 64 | 0 | 64
    100 | 18 |  | 18
    90: number analyzed (Participants) | 64 | 0 | 64
    90 | 28 |  | 28
    80: number analyzed (Participants) | 64 | 0 | 64
    80 | 13 |  | 13
    70: number analyzed (Participants) | 64 | 0 | 64
    70 | 2 |  | 2
    60: number analyzed (Participants) | 64 | 0 | 64
    60 | 1 |  | 1
    50: number analyzed (Participants) | 64 | 0 | 64
    50 | 2 |  | 2
    less than 50: number analyzed (Participants) | 64 | 0 | 64
    less than 50 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Remission Rate (ORR) Per Independent Review Committee (IRC) (for ALL Participants)
Description: ORR is defined as the percentage of participants with a best overall disease response of complete remission (CR) or Complete remission with incomplete blood count recovery (CRi), where the best overall disease response is defined as the best disease response recorded from CTL019 infusion until the start of new anticancer therapy. Best response was assigned in the following order: CR, CRi, CR or CRi with residual mediastinal disease, No response and Unknown.
Time Frame: within 6 months after CTL019 infusion
Population: Efficacy Analysis Set (EAS): A subset of all infused patients who were treated with CTL019 at least 6 months prior to the clinical data cutoff. In the final analysis, it is identical to the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - All Participants
Number analyzed (Participants) | 64
Percentage of participants | 70.3 [57.6 to 81.1]
Statistical Analysis 1: Comparison: Tisagenlecleucel (CTL019) - All Participants; Test type: Other; p < 0.0001, Clopper-Pearson

2. Primary Outcome: Overall Remission Rate (ORR) Per Local Investigator Assessment (for Lymphoblastic Lymphoma Patients Only)
Description: Overall Remission Rate (ORR), which includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi), as determined by assessments of peripheral blood, bone marrow, CNS symptoms, physical exam (PE) and cerebrospinal fluid (CSF). This primary endpoint was based on the local investigator assessment. No participants with lymphoblastic lymphoma were infused in this study.
Time Frame: 6 months after CTL019
Population: Efficacy Analysis Set (EAS): A subset of all infused patients who were treated with CTL019 at least 6 months prior to the clinical data cutoff. In the final analysis, it is identical to the FAS. No patients with Lymphoblastic Lymphoma were enrolled in this trial, hence there is no data to report.
Groups:
- Tisagenlecleucel (CTL019) - Local Assessment: Pediatric participants with r/r B-cell ALL
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With Clinical Response Without Stem Cell Transplantation (SCT) at Month 6 - Per IRC Assessment
Description: Evaluate the percentage of participants who achieved CR or CRi at Month 6 without SCT between tisagenlecleucel infusion and Month 6 response assessment.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tisagenlecleucel (CTL019) - IRC Assessment: Pediatric participants with r/r B-cell ALL
Arm/Group | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 64
Percentage of participants | 53.1 [40.2 to 65.7]

4. Secondary Outcome: Percentage of Subjects Who Achieved CR or CRi and Then Proceeded to SCT While in Remission Prior to Month 6 Response - Per IRC Assessment
Description: Evaluate the percentage of subjects who achieved CR or CRi and then proceeded to SCT while in remission prior to Month 6 response assessment.
Time Frame: prior to Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tisagenlecleucel (CTL019) - Per IRC Assessment: Pediatric participants with r/r B-cell ALL
Arm/Group | Tisagenlecleucel (CTL019) - Per IRC Assessment
Number analyzed (Participants) | 64
Percentage of participants | 7.8 [2.6 to 17.3]

5. Secondary Outcome: Duration of Remission (DOR) Per Local and IRC Assessment
Description: DOR is the time from achievement of CR or CRi, whichever occurs first, to relapse or death due to ALL
Time Frame: From CR or CRi to relapse or death up to 60 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 64 | 64
months | NA [13.6 to NA] — N/A = median DOR was not reached as there were not enough participants with DOR events | NA [13.6 to NA] — N/A = median DOR was not reached as there were not enough participants with DOR events

6. Secondary Outcome: Percentage of Participants With CR or CRi With Minimum Residual Disease (MRD) Negative Bone Marrow 6 Months After CTL019 Infusion
Description: Percentage of participants with best overall response (BOR) of CR or CRi with MRD negative bone marrow status 6 months after CTL019 infusion among all participants who achieved CR or CRi per Local Investigator & IRC assessment
Time Frame: within 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 64 | 64
Percentage of participants | 67.2 [54.3 to 78.4] | 67.2 [54.3 to 78.4]

7. Secondary Outcome: Relapse-free Survival (RFS) for Responders Per Local and IRC Assessment
Description: RFS is the time from achievement of CR or CRi whichever occurs first to relapse or death due to any cause during CR or CRi.
Time Frame: 60 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 45 | 45
months | NA [13.6 to NA] — N/A = median RFS was not reached as there were not enough participants with RFS events | NA [13.6 to NA] — N/A = median RFS was not reached as there were not enough participants with RFS events

8. Secondary Outcome: Event-free Survival (EFS) Per Local and IRC Assessment
Description: EFS is the time from date of CTL019 infusion to the earliest of death, relapse or treatment failure. Treatment failure is defined as "no response" in the study and discontinuation from the study due to any of the following reasons: death, AE, lack of efficacy, new anticancer therapy.
Time Frame: 60 Months
Population: FAS: All subjects who received an infusion of CTL019
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 64 | 64
months | 15.6 [6.4 to NA] — N/A = not estimable because there were not enough participants who had an EFS event to estimate the upper limit of the median EFS | 15.6 [6.4 to NA] — N/A = not estimable because there were not enough participants who had an EFS event to estimate the upper limit of the median EFS

9. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from date of CTL019 infusion to the date of death due to any reason
Time Frame: 60 Months
Population: FAS: All subjects who received an infusion of CTL019
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - All Participants
Number analyzed (Participants) | 64
months | 29.9 [15.1 to 42.4]

10. Secondary Outcome: Secondary Outcome: Percentage of Participants Attaining CR or CRi With MRD Negative Bone Marrow Status at Day 28 +/- 4 Days After CTL019 Infusion
Description: Percentage of participants attaining CR or CRi with MRD negative bone marrow status at Day 28 +/- 4 days after CTL019 infusion per Local Investigator and IRC assessment. BM MRD were only collected and measured only within responders.
Time Frame: Day 28
Population: Efficacy Analysis Set (EAS): A subset of all infused patients who were treated with CTL019 at least 6 months prior to the clinical data cutoff. In the final analysis, it is identical to the FAS. BM MRD were only collected and measured only within responders.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 64 | 64
Percentage of participants
  With BM MRD -ve: i.e. MRD% < 0.01% | 71.9 [59.2 to 82.4] | 71.9 [59.2 to 82.4]
  With BM 0.01% <= MRD% < 5% | 1.6 [NA to NA] — N/A: only 1 participant with BM MRD to calculate meaningful confidence interval (CI) | 1.6 [NA to NA] — N/A: only 1 participant with BM MRD to calculate meaningful confidence interval (CI)
  With BM MRD% >= 5% | 1.6 [NA to NA] — N/A: only 1 participant with BM MRD to calculate meaningful CI | 1.6 [NA to NA] — N/A: only 1 participant with BM MRD to calculate meaningful CI
  BM MRD not available | 6.3 [NA to NA] — N/A: few participants with BM MRD to provide meaningful CI | 6.3 [NA to NA] — N/A: few participants with BM MRD to provide meaningful CI

11. Secondary Outcome: CTL019 Transgene Levels by qPCR CTL019 Cells by in qPCR Blood and Bone Marrow
Description: Characterize the in vivo cellular pharmacokinetic (PK) profile (levels,persistence, trafficking) of CTL019 cells in target tissues
Time Frame: Enrollment; D1; D4; D7; D11; D14; D21; D28; M3; M6; M9, M12; M18; M24, M30, M36, M42, M48 for transgene levels in blood; Screening, D28, M3, M6 for transgene levels in bone marrow
Population: Pharmacokinetic Analysis Set (PAS): A subset of FAS who have at least one sample providing evaluable pharmacokinetic (PK) data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug DNA
Groups:
- CR/CRi: Participants had Complete remission (CR)/Complete remission with incomplete blood count recovery (CRi)
- No Response (NR): No response was defined as failure to attain the criteria needed for any response categories or relapse
- Unknown: unknown was assigned in case the baseline assessment or the response assessment was not done, incomplete, indeterminate or not performed within the respective time frame.
Arm/Group | CR/CRi | No Response (NR) | Unknown
Number analyzed (Participants) | 52 | 6 | 6
copies/ug DNA
  Enrollment blood: number analyzed (Participants) | 49 | 6 | 5
  Enrollment blood | NA (NA) — N/A: No CTL019 was infused at the enrollment | NA (NA) — N/A: No CTL019 was infused at the enrollment | NA (NA) — N/A: No CTL019 was infused at the enrollment
  Day 1 (D1): blood: number analyzed (Participants) | 41 | 4 | 6
  Day 1 (D1): blood | 3680 (344.3) | 3190 (348.6) | 2440 (220.6)
  D4: blood: number analyzed (Participants) | 48 | 6 | 6
  D4: blood | 234 (197.8) | 48.8 (282.4) | 88.0 (71.0)
  D7: blood: number analyzed (Participants) | 51 | 6 | 6
  D7: blood | 4460 (616.2) | 231 (499.1) | 402 (114.7)
  D11: blood: number analyzed (Participants) | 34 | 4 | 4
  D11: blood | 21200 (262.3) | 423 (52.7) | 1920 (8318.1)
  D14: blood: number analyzed (Participants) | 49 | 6 | 5
  D14: blood | 12500 (292.1) | 1600 (337.1) | 42835.8 (9060)
  D21: blood: number analyzed (Participants) | 49 | 6 | 5
  D21: blood | 3720 (480.5) | 7750 (334.5) | 1050 (220743.9)
  D28: blood: number analyzed (Participants) | 52 | 6 | 3
  D28: blood | 1360 (650.3) | 2770 (684.8) | 515 (244650713.9)
  Month 3 (M3): blood: number analyzed (Participants) | 49 | 2 | 2
  Month 3 (M3): blood | 220 (224.3) | 690 (NA) — N/A = not estimable because too few participants to calculate Geometric CV | 564 (NA) — N/A = not estimable because too few participants to calculate Geometric CV
  Month M6: blood: number analyzed (Participants) | 40 | 1 | 1
  Month M6: blood | 146 (157.5) | NA (NA) — N/A = not estimable because too few participants to calculate Geometric CV; also, the geometric mean was not applicable for NR group at Month 6 as the arithmetic mean was zero | 127 (NA) — N/A = not estimable because too few participants to calculate Geometric CV
  Month M9: blood: number analyzed (Participants) | 30 | 0 | 0
  Month M9: blood | 117 (179.3) |  |
  Month M12: blood: number analyzed (Participants) | 30 | 0 | 0
  Month M12: blood | 113 (312.4) |  |
  Month M18: blood: number analyzed (Participants) | 18 | 0 | 0
  Month M18: blood | 87.2 (200.3) |  |
  Month M24: blood: number analyzed (Participants) | 15 | 0 | 0
  Month M24: blood | 92.7 (160.5) |  |
  Month M30: blood: number analyzed (Participants) | 5 | 0 | 0
  Month M30: blood | 59.9 (150.0) |  |
  Month M36: blood: number analyzed (Participants) | 3 | 0 | 0
  Month M36: blood | 10.7 (19.9) |  |
  Month M42: blood: number analyzed (Participants) | 2 | 0 | 0
  Month M42: blood | 35.3 (NA) — N/A = not estimable because too few participants to calculate Geometric CV |  |
  Month M48: blood: number analyzed (Participants) | 1 | 0 | 0
  Month M48: blood | NA (NA) — NA = geometric mean is not estimable because the CTL019 transgene level for the only one patient is 0. |  |
  Screening: Bone marrow (BM): number analyzed (Participants) | 47 | 6 | 6
  Screening: Bone marrow (BM) | NA (NA) — N/A = No CTL019 was infused at screening | NA (NA) — N/A = No CTL019 was infused at screening | NA (NA) — N/A = No CTL019 was infused at screening
  D28 BM: number analyzed (Participants) | 50 | 4 | 4
  D28 BM | 646 (1009.7) | 969 (166.8) | 615 (4763885.9)
  M3 BM: number analyzed (Participants) | 40 | 0 | 2
  M3 BM | 179 (182.5) |  | 542 (NA) — N/A = not estimable because too few participants to calculate Geometric CV
  M6 BM: number analyzed (Participants) | 32 | 1 | 0
  M6 BM | 133 (121.7) | 35.3 (NA) — N/A = not estimable because too few participants to calculate Geometric CV |

12. Secondary Outcome: Humoral Immunogenicity Interpretation by Day 28 Disease Response Per IRC (Anti-CTL019 Antibodies)
Description: Humoral immunogenicity was measured by anti-CTL019 antibodies in human serum using a flow cytometry method. (Prevalence and incidence of immunogenicity to CTL019)
Time Frame: Baseline; Day 14; Day 28; Month 3; Month 6; Month 12; Month 24, Month 36
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Number; unit: Percentage of participants
Groups:
- No Response: No response was defined as failure to attain the criteria needed for any response categories or relapse
Arm/Group | CR/CRi | No Response | Unknown
Number analyzed (Participants) | 52 | 6 | 6
Percentage of participants
  Baseline: Positive | 67.3 | 66.7 | 83.3
  Day 14: Positive | 84.6 | 100 | 83.3
  Day 28: Positive | 80.8 | 100 | 50.0
  Month 3: Positive | 75.0 | 16.7 | 33.3
  Month 6: Positive | 63.5 | 16.7 | 16.7
  Month 12: Positive | 46.2 | 0 | 0
  Month 24: Positive | 11.5 | 0 | 0
  Month 36: Positive | 9.6 | 0 | 0

13. Secondary Outcome: ORR by Low Baseline Bone Marrow Burden Within 6 Months Post CTL019 Infusion
Description: ORR within 6 months after infusion of CTL019 per Local & IRC assessment by baseline bone marrow tumor burden presence.
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 12 having a low bone marrow tumor burden at enrollment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 12 | 12
percentage of participants | 83.3 [51.6 to 97.9] | 83.3 [51.6 to 97.9]

14. Secondary Outcome: ORR by High Baseline Bone Marrow Burden Within 6 Months Post CTL019 Infusion
Description: ORR within 6 months after infusion of CTL019 per Local Investigator & IRC assessment by high baseline bone marrow tumor burden presence.
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 30 having a high bone marrow tumor burden at enrollment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 30 | 30
percentage of participants | 63.3 [43.9 to 80.1] | 63.3 [43.9 to 80.1]

15. Secondary Outcome: ORR by Baseline Extramedullary Disease Presence of Yes Within 6 Months Post CTL019 Infusion
Description: ORR within 6 months after infusion of CTL019 per Local Investigator & IRC assessment by baseline extramedullary disease presence of Yes.
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 2 participants having a baseline extramedullary presence.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 2 | 2
percentage of participants | 100 [NA to NA] — N/A: no confidence interval for 100% response | 100 [NA to NA] — N/A: no confidence interval for 100% response

16. Secondary Outcome: ORR by Baseline Extramedullary Disease Presence of No Within 6 Months Post CTL019 Infusion
Description: ORR within 6 months after infusion of CTL019 per Local Investigator & IRC assessment by baseline extramedullary disease presence of No.
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 40 participants having no baseline extramedullary presence.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 40 | 40
percentage of participants | 67.5 [50.9 to 81.4] | 67.5 [50.9 to 81.4]

17. Secondary Outcome: Bone Marrow (BM) Minimum Residual Disease (MRD) Status by Flow Cytometry Within 6 Months Post CTL019 Infusion by High Baseline Bone Marrow Tumor Burden
Description: BM MRD status was by Local Investigator and IRC assessment within 6 months after infusion of CTL019 by baseline bone marrow tumor burden. BM MRD were collected and measured only within responders.
Time Frame: Within 6 months
Population: Efficacy Analysis Set: A subset of FAS treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on cut-off date of 6-Oct-2017, with only 42 participants and 30 having a high baseline bone marrow tumor burden. BM MRD were collected and measured only within responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 30 | 30
percentage of participants
  Had BOR of CR/CRi with BM MRD -ve (MRD%< 0.01%) | 56.7 [37.4 to 74.5] | 56.7 [37.4 to 74.5]
  Had BOR of CR/CRi with BM 0.01% <= MRD% < 5% | 6.7 [NA to NA] — N/A = too few participants to calculate a meaningful CI | 6.7 [NA to NA] — N/A = too few participants to calculate a meaningful CI

18. Secondary Outcome: Bone Marrow MRD Status Was by Flow Cytometry Within 6 Months Post CTL019 Infusion by Low Baseline Bone Marrow Tumor Burden
Description: BM MRD status was per Local Investigator and IRC assessment within 6 months after infusion of CTL019 by low baseline bone marrow tumor burden. BM MRD were collected and measured only within responders.
Time Frame: Within 6 months
Population: Efficacy Analysis Set: A subset of FAS treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on cut-off date of 6-Oct-2017, with only 42 participants and 12 having a high baseline bone marrow tumor burden. BM MRD were collected and measured only within responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 12 | 12
percentage of participants | 83.3 [51.6 to 97.9] | 83.3 [51.6 to 97.9]

19. Secondary Outcome: Bone Marrow MRD Status by Flow Cytometry Within 6 Months Post CTL019 Infusion by Baseline Extramedullary Disease Presence: Yes
Description: BM MRD status was by Local Investigator and IRC assessment within 6 months after infusion pf CTL019 by baseline extramedullary disease presence of Yes. BM MRD were collected and measured only within responders.
Time Frame: Within 6 months
Population: Efficacy Analysis Set: A subset of FAS treated with CTL019 at least 6 months prior to the clinical data cutoff. FAS: All subjects who received an infusion of CTL019. Data is based on cut-off date of 6-Oct-2017, with only 42 participants & 2 having a BL extramedullary disease presence of Yes. BM MRD were collected & measured only within responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 2 | 2
percentage of participants | 100 [15.8 to 100] | 100 [15.8 to 100]

20. Secondary Outcome: Bone Marrow MRD Status by Flow Cytometry Within 6 Months Post CTL019 Infusion by Baseline Extramedullary Disease Presence: No
Description: BM MRD status WAS per Local Investigator and IRC assessment within 6 months after infusion pf CTL019 by baseline extramedullary disease presence of No. BM MRD were collected and measured only within responders.
Time Frame: Within 6 months
Population: Efficacy Analysis Set: A subset of FAS treated with CTL019 at least 6 months prior to the clinical data cutoff. FAS: All subjects who received an infusion of CTL019. Data is based on cut-off date of 6-Oct-2017, with only 42 participants & 40 having a BL extramedullary disease presence of No. BM MRD were collected & measured only within responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 40 | 40
percentage of participants
  With BM MRD -ve (MRD%< 0.01%) | 62.5 [45.8 to 77.3] | 62.5 [45.8 to 77.3]
  With bone marrow 0.01% <= MRD% < 5% | 5.0 [NA to NA] — N/A = too few participants to calculate CI | 5.0 [NA to NA] — N/A = too few participants to calculate CI

21. Secondary Outcome: Duration of Remission (DoR) Censoring Hematopoietic Stem Cell Transplantation (HSCT) by Low Baseline Bone Marrow Tumor Burden
Description: DoR per Local Investigator & IRC assessment by low baseline marrow tumor burden
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 12 having a low baseline marrow tumor burden
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 12 | 12
months | NA [5.4 to NA] — N/A = median DoR was not reached as there were not enough participants with DoR events | NA [5.4 to NA] — N/A = median DoR was not reached as there were not enough participants with DoR events

22. Secondary Outcome: Duration of Remission (DoR) Censoring HSCT by High Baseline Bone Marrow Tumor Burden
Description: DoR per Local Investigator & IRC assessment by high baseline bone marrow tumor burden
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 30 having a high baseline marrow tumor burden
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 30 | 30
months | NA [5.3 to NA] — N/A = median DoR was not reached as there were not enough participants with DoR events | NA [5.3 to NA] — N/A = median DoR was not reached as there were not enough participants with DoR events

23. Secondary Outcome: Duration of Remission (DoR) Censoring HSCT by Baseline Extramedullary Disease Presence: Yes
Description: DoR per Local Investigator & IRC assessment by baseline extramedullary disease presence of Yes.
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 2 having a baseline extramedullary disease presence of Yes
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 2 | 2
months | NA [3.4 to NA] — N/A = median DoR was not reached as there were not enough participants with D0R events | NA [3.4 to NA] — N/A = median DoR was not reached as there were not enough participants with DoR events

24. Secondary Outcome: Duration of Remission (DoR) Censoring HSCT by Baseline Extramedullary Disease Presence: No
Description: DoR per Local Investigator & IRC assessment by baseline extramedullary disease presence of No
Time Frame: Within 6 months
Population: EAS: Efficacy Analysis Set (EAS): A subset of full analysis set (FAS) who were treated with CTL019 at least 6 months prior to the clinical data cutoff FAS: All subjects who received an infusion of CTL019. Data is based on data cut-off date of 6-Oct-2017, with only 42 participants and 40 having a baseline extramedullary disease presence of No
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel (CTL019) - Local Assessment | Tisagenlecleucel (CTL019) - IRC Assessment
Number analyzed (Participants) | 40 | 40
months | NA [5.9 to NA] — N/A = median DOR was not reached as there were not enough participants with DOR events | NA [5.9 to NA] — N/A = median DOR was not reached as there were not enough participants with DOR events

25. Secondary Outcome: Participants Achieving Cellular Immunogenicity Net Response by Day 28 Response Per IRC
Description: Activation of T cells in PBMC collected from subjects in response to mCAR19 -derived peptides was used to assess the cellular immunogenicity against tisagenlecleucel. CD4 and CD8 T cell net responses (in %) were calculated for 2 non-overlapping CTL019 peptide pools (i.e., Pool 1 and Pool 2). (Lymphocyte subsets of B and T cells and description of associated safety events)
Time Frame: Baseline; Day 14; Day 28; Month 3; Month 6; Month 12; Month 24, Month 36
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Number; unit: Percentage of participants
Arm/Group | CR/CRi | No Response | Unknown
Number analyzed (Participants) | 52 | 6 | 6
Percentage of participants
  Baseline: Pool 1 CD3+ CD4+ IFNg+ | 92.3 | 83.3 | 50.0
  Day 14: Pool 1 CD3+ CD4+ IFNg+ | 82.7 | 100 | 50.0
  Day 28: Pool 1 CD3+ CD4+ IFNg+ | 94.2 | 100 | 50.0
  Month 3: Pool 1 CD3+ CD4+ IFNg+ | 82.7 | 16.7 | 33.3
  Month 6: Pool 1 CD3+ CD4+ IFNg+ | 67.3 | 16.7 | 57.8
  Month 12: Pool 1 CD3+ CD4+ IFNg+ | 48.1 | 0 | 0
  Month 24: Pool 1 CD3+ CD4+ IFNg+ | 17.3 | 0 | 0
  Month 36: Pool 1 CD3+ CD4+ IFNg+ | 9.6 | 0 | 0
  Baseline: Pool 2 CD3+ CD4+ IFNg+ | 92.3 | 83.3 | 50.0
  Day 14: Pool 2 CD3+ CD4+ IFNg+ | 82.7 | 100 | 50.0
  Day 28: Pool 2 CD3+ CD4+ IFNg+ ) | 94.2 | 100 | 50.0
  Month 3: Pool 2 CD3+ CD4+ IFNg+ | 82.7 | 16.7 | 33.3
  Month 6: Pool 2 CD3+ CD4+ IFNg+ | 67.3 | 16.7 | 16.7
  Month 12: Pool 2 CD3+ CD4+ IFNg+ | 48.1 | 0 | 0
  Month 24: Pool 2 CD3+ CD4+ IFNg+ | 17.3 | 0 | 0
  Month 36: Pool 2 CD3+ CD4+ IFNg+ | 9.6 | 0 | 0
  Baseline: Pool 1 CD3+ CD8+ IFNg+ | 92.3 | 83.3 | 50.0
  Day 14: Pool 1 CD3+ CD8+ IFNg+ | 82.7 | 100 | 50.0
  Day 28: Pool 1 CD3+ CD8+ IFNg+: number analyzed (Participants) | 41 | 6 | 2
  Day 28: Pool 1 CD3+ CD8+ IFNg+ | 94.2 | 100 | 50.0
  Month 3: Pool 1 CD3+ CD8+ IFNg+ | 82.7 | 16.7 | 33.3
  Month 6: Pool 1 CD3+ CD8+ IFNg+ | 67.3 | 16.7 | 16.7
  Month 12: Pool 1 CD3+ CD8+ IFNg+ | 48.1 | 0 | 0
  Month 24: Pool 1 CD3+ CD8+ IFNg+ | 17.3 | 0 | 0
  Month 36: Pool 1 CD3+ CD8+ IFNg+ | 9.6 | 0 | 0
  Baseline: Pool 2 CD3+ CD8+ IFNg+ | 92.3 | 83.3 | 50.0
  Day 14: Pool 2 CD3+ CD8+ IFNg+ | 82.7 | 100 | 50.0
  Day 28: Pool 2 CD3+ CD8+ IFNg+ | 94.2 | 100 | 50.0
  Month 3: Pool 2 CD3+ CD8+ IFNg+ | 82.7 | 16.7 | 33.3
  Month 6: Pool 2 CD3+ CD8+ IFNg+ | 67.3 | 16.7 | 16.7
  Month 12: Pool 2 CD3+ CD8+ IFNg+ | 48.1 | 0 | 0
  Month 24: Pool 2 CD3+ CD8+ IFNg+ | 17.3 | 0 | 0
  Month 36: Pool 2 CD3+ CD8+ IFNg+ | 9.6 | 0 | 0

26. Secondary Outcome: Peripheral Blood PK Parameters for Tisagenlecleucel Transgene Levels by qPCR, by Day 28 Disease Response by Local & IRC Assessment: AUC0-28d and AUC0-84d
Description: Characterize the in vivo cellular pharmacokinetic (PK) profile. AUC0-28d and AUC0-84d is defined as the AUC from time zero to day 28 and 84 or other disease assessment days, in peripheral blood (% or copies/μg x days). Data was only reported for evaluable PK parameters. The Overall Number of Participants Analyzed represents all participants for which a baseline assessment was collected for this Outcome Measure, and therefore these participants did contribute data to this estimation parameter, whereas the Number Analyzed per Row represents the number of participants with data available at either 28 or 84 days.
Time Frame: 0 - 28 days post-infusion for AUC0-28d and 0 - 84 days post-infusion for AUC0-84d
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/µg*days
Arm/Group | CR/CRi | No Response (NR) | Unknown
Number analyzed (Participants) | 52 | 6 | 6
copies/µg*days
  AUC0-28d: number analyzed (Participants) | 52 | 3 | 1
  AUC0-28d | 261000 (199.8) | 151000 (71.7) | 617000 (NA) — N/A = Too few participants to calculate geometric CV
  AUC0-84d: number analyzed (Participants) | 45 | 2 | 1
  AUC0-84d | 368000 (182.9) | 443000 (79.9) | 1340000 (NA) — N/A = Too few participants to calculate geometric CV

27. Secondary Outcome: Peripheral Blood PK Parameters for Tisagenlecleucel Transgene Levels by qPCR, by Day 28 Disease Response by Local & IRC Assessment: Cmax
Description: Characterize the in vivo cellular pharmacokinetic (PK) profile. Cmax is defined as the maximum (peak) observed in peripheral blood drug concentration after single dose administration (% or copies/μg).
Time Frame: Day 28
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/µg
Arm/Group | CR/CRi | No Response (NR) | Unknown
Number analyzed (Participants) | 52 | 5 | 3
copies/µg | 28300 (197.0) | 15100 (49.4) | 52500 (91.1)

28. Secondary Outcome: Peripheral Blood PK Parameters for Tisagenlecleucel Transgene Levels by qPCR, by Day 28 Disease Response by Local & IRC Assessment: Tmax
Description: Characterize the in vivo cellular pharmacokinetic (PK) profile. Tmax is defined as the time to reach maximum (peak) peripheral blood drug concentration after single dose administration (days)
Time Frame: Day 28
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | CR/CRi | No Response (NR) | Unknown
Number analyzed (Participants) | 52 | 5 | 2
days | 9.84 [6.74 to 54.8] | 20.0 [13.9 to 22.8] | 11.9 [11.0 to 12.9]

29. Secondary Outcome: Peripheral Blood PK Parameters for Tisagenlecleucel Transgene Levels by qPCR, by Day 28 Disease Response by Local & IRC Assessment: T1/2
Description: Characterize the in vivo cellular pharmacokinetic (PK) profile. T1/2 is defined as the half-life associated with the disposition phase slopes (alpha, beta, gamma etc.) of a semi logarithmic concentration-time curve (days) in peripheral blood
Time Frame: Day 28
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | CR/CRi | No Response (NR) | Unknown
Number analyzed (Participants) | 34 | 2 | 1
days | 31.9 (415.1) | 4.36 (421.2) | 42.1 (NA) — N/A = with only 1 subject, geometric CV could not be calculated

30. Secondary Outcome: Peripheral Blood PK Parameters for Tisagenlecleucel Transgene Levels by qPCR, by Day 28 Disease Response by Local & IRC Assessment: Clast
Description: Characterize the in vivo cellular pharmacokinetic (PK) profile. Clast is defined as the last observed quantifiable concentration in peripheral blood (% or copies/ug)
Time Frame: Day 28
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/µg
Arm/Group | CR/CRi | No Response (NR) | Unknown
Number analyzed (Participants) | 52 | 5 | 1
copies/µg | 223 (283.4) | 1980 (207.5) | 80.3 (NA) — N/A = with only 1 subject, geometric CV could not be calculated

31. Secondary Outcome: Peripheral Blood PK Parameters for Tisagenlecleucel Transgene Levels by qPCR, by Day 28 Disease Response by Local & IRC Assessment: Tlast
Description: Characterize the in vivo cellular pharmacokinetic (PK) profile. Tlast is defined as the time of last observed quantifiable concentration in peripheral blood (days)"
Time Frame: Day 28
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | CR/CRi | No Response (NR) | Unknown
Number analyzed (Participants) | 52 | 5 | 1
days | 179 [17.8 to 921] | 26.9 [26.7 to 96.1] | 210 [210 to 210]

32. Secondary Outcome: CD19 Status of Bone Marrow/Blood Relapse in FAS Patients Who Achieved CR or CRi and Then Relapsed
Description: The CD19 status of bone marrow/blood relapse was categorized as follows: CD19 positive, CD19 dim, CD19 negative, CD19 positive/negative & CD19 unknown
Time Frame: At time of relapse up to 60 months
Population: FAS patients who achieved CR & CRi and then relapsed. FAS: All subjects who received an infusion of CTL019
Measure: Number; unit: Percentage of participants
Groups:
- Tisagenlecleucel - FAS Pts Who Achieved CR/CRi & Then Relapsed: Pediatric participants with r/r B-cell who were infused with tisagenlecleucel and then relapsed
Arm/Group | Tisagenlecleucel - FAS Pts Who Achieved CR/CRi & Then Relapsed
Number analyzed (Participants) | 21
Percentage of participants
  CD19 status of BM/blood relapse:positive | 22.2
  CD19 status of BM/blood relapse: dim | 5.6
  CD19 status of BM/blood relapse: negative | 16.7
  CD19 status of BM/blood relapse: +ve/-ve | 16.7
  CD19 status of BM/blood relapse: Unknown | 55.6

33. Secondary Outcome: Site of Initial Relapse Among FAS Patients Who Achieved CR/CRi and Then Relapsed
Description: This is the site of involvement of initial relapse after achieving a best overall response of CR/CRi.
Time Frame: At time of relapse up to 60 months
Population: FAS patients who achieved CR & CRi and then relapsed. FAS: All subjects who received an infusion of CTL019
Measure: Number; unit: Percentage of participants
Arm/Group | Tisagenlecleucel - FAS Pts Who Achieved CR/CRi & Then Relapsed
Number analyzed (Participants) | 21
Percentage of participants
  BM/blood relapse | 72.2
  Extramedullary only | 27.8
  Unknown | 16.7

34. Secondary Outcome: Time to B-cell Recovery in Participants Who Achieved CR or CRi by IRC
Description: Time to B cell recovery was defined as the time from onset of remission to the earliest time when the percentage of CD19+ total B cell among viable WBC is ≥ 1% or among lymphocyte is at least 3%.
Time Frame: during the whole study, up to 60 months
Population: FAS patients who achieved CR or CRi. FAS: All subjects who received an infusion of CTL019
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisagenlecleucel (CTL019) - All Participants
Number analyzed (Participants) | 54
Months | 35.5 [7.6 to NA] — N/A = not estimable because there were not enough participants who had events to estimate the upper limit of the median

35. Secondary Outcome: Percentage of CD19+ B Cell Levels in Peripheral Blood by Day 28 Disease Response by IRC Assessment
Description: The levels (%) of CD19+ total B cells amongst viable white blood cells (WBC) in peripheral blood
Time Frame: Enrollment/Pre-Chemotherapy; Pre-infusion; Baseline; Day 7; Day 14; Day 21; Day 28; Month 3; Month 6; Month 9; Month 12; Month 24; Month 36
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Mean (Standard Deviation); unit: Percentage of CD19+ B cell levels
Arm/Group | CR/CRi | No Response | Unknown
Number analyzed (Participants) | 52 | 6 | 6
Percentage of CD19+ B cell levels
  Enrollment/Pre-Chemotherapy: number analyzed (Participants) | 50 | 6 | 6
  Enrollment/Pre-Chemotherapy | 26.8 (28.733) | 52.29 (36.758) | 32.66 (28.102)
  Pre-infusion: number analyzed (Participants) | 1 | 0 | 1
  Pre-infusion | 0.02 (NA) — N/A = Too few participants to calculate geometric SD |  | 46.80 (NA) — N/A = Too few participants to calculate geometric SD
  Baseline: number analyzed (Participants) | 50 | 6 | 6
  Baseline | 25.11 (28.584) | 52.29 (36.758) | 29.50 (24.466)
  Day 7: number analyzed (Participants) | 45 | 6 | 6
  Day 7 | 1.06 (3.735) | 34.40 (46.922) | 23.18 (38.772)
  Day 14: number analyzed (Participants) | 50 | 6 | 5
  Day 14 | 0.73 (5.096) | 33.76 (45.359) | 3.43 (7.520)
  Day 21: number analyzed (Participants) | 46 | 6 | 5
  Day 21 | 0.01 (0.017) | 19.67 (32.553) | 16.13 (35.929)
  Day 28: number analyzed (Participants) | 48 | 6 | 3
  Day 28 | 0.02 (0.069) | 34.97 (36.648) | 0.02 (0.012)
  Month 3: number analyzed (Participants) | 44 | 1 | 2
  Month 3 | 0.79 (1.971) | 0.57 (NA) — N/A = Too few participants to calculate geometric SD | 11.26 (15.917)
  Month 6: number analyzed (Participants) | 37 | 1 | 1
  Month 6 | 1.86 (7.958) | 9.70 (NA) — N/A = Too few participants to calculate geometric SD | 0.01 (NA) — N/A = Too few participants to calculate geometric SD
  Month 9: number analyzed (Participants) | 27 | 0 | 0
  Month 9 | 0.63 (2.180) |  |
  Month 12: number analyzed (Participants) | 27 | 0 | 0
  Month 12 | 0.85 (2.420) |  |
  Month 24: number analyzed (Participants) | 14 | 0 | 0
  Month 24 | 1.74 (3.446) |  |
  Month 36: number analyzed (Participants) | 6 | 0 | 0
  Month 36 | 1.10 (2.106) |  |

36. Secondary Outcome: Key Inflammatory Markers and Cytokine Parameters in Blood Within 1 Month by Maximum Cytokine Release Syndrome (CRS) Grade: C Reactive Protein (CRP)
Description: C-Reactive Protein at Pre-infusion, baseline, and change from baseline for Days 7, 14, 21, 28, Month 3
Time Frame: Pre-infusion, Baseline, Day 7, Day 14, Day 21, Day 28, Month 3
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Median (Full Range); unit: mg/L
Groups:
- NO CRS: No cytokine release syndrome
- Grade 1/2: Grade 1 and 2 of cytokine release syndrome post tisagenlecleucel infusion
- Grade 3: Grade 3 of cytokine release syndrome post tisagenlecleucel infusion
- Grade 4: Grade 4 of cytokine release syndrome post tisagenlecleucel infusion
- All Participants: All participants with & without CRS
Arm/Group | NO CRS | Grade 1/2 | Grade 3 | Grade 4 | All Participants
Number analyzed (Participants) | 14 | 31 | 8 | 11 | 64
mg/L
  Pre-infusion: number analyzed (Participants) | 14 | 29 | 8 | 9 | 60
  Pre-infusion | 9.21 [2.9 to 34.0] | 8.27 [2.0 to 1530.0] | 7.45 [0.6 to 50.0] | 9.00 [2.0 to 153.0] | 9.00 [0.6 to 1530.0]
  Baseline (BL): number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Baseline (BL) | 9.21 [2.9 to 34.0] | 9.04 [2.0 to 1530.0] | 7.45 [0.6 to 50.0] | 9.00 [2.0 to 153.0] | 9.00 [0.6 to 1530.0]
  Change from BL Day7: number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Change from BL Day7 | 0.00 [-15.0 to 25.0] | 15.00 [-460.0 to 215.0] | 79.55 [-2.0 to 380.0] | 108.00 [-125.0 to 255.0] | 9.10 [-460.0 to 380.0]
  Change from BL Day 14: number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Change from BL Day 14 | 0.00 [-20.0 to 24.0] | 0.00 [-1031.0 to 215.0] | 10.50 [-42.0 to 199.0] | 15.70 [-148.0 to 100.0] | 0.00 [-1031.0 to 215.0]
  Change from BL Day 21: number analyzed (Participants) | 14 | 28 | 8 | 7 | 57
  Change from BL Day 21 | 0.00 [-14.0 to 29.5] | -0.80 [-1460.0 to 677.0] | 2.00 [-42.0 to 37.0] | -3.00 [-57.0 to 73.0] | 0.00 [-1460.0 to 677.0]
  Change from BL Day 28: number analyzed (Participants) | 14 | 27 | 8 | 9 | 59
  Change from BL Day 28 | 0.00 [-15.0 to 47.0] | -0.70 [-1487.0 to 47.0] | 1.50 [-45.0 to 55.0] | -3.00 [-151.0 to 27.0] | 0.00 [-1487.0 to 55.0]
  Change from BL Month 3: number analyzed (Participants) | 11 | 23 | 5 | 7 | 46
  Change from BL Month 3 | 0.00 [-12.1 to 101.0] | -1.00 [-1501.0 to 7.1] | 0.00 [-3.0 to 120.5] | -1.00 [-149.0 to 13.0] | -0.65 [-1501.0 to 120.5]

37. Secondary Outcome: Key Inflammatory Markers and Cytokine Parameters in Blood Within 1 Month by Maximum Cytokine Release Syndrome (CRS) Grade: Ferritin
Description: Ferritin at Pre-infusion, baseline, and change from baseline for Days 7, 14, 21, 28, Month 3
Time Frame: Pre-infusion, Baseline, Day 7, Day 14, Day 21, Day 28, Month 3
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Median (Full Range); unit: ug/L
Arm/Group | NO CRS | Grade 1/2 | Grade 3 | Grade 4 | All Participants
Number analyzed (Participants) | 14 | 31 | 8 | 11 | 64
ug/L
  Pre-infusion: number analyzed (Participants) | 14 | 26 | 8 | 9 | 54
  Pre-infusion | 1865.20 [459.0 to 5015.0] | 2202.22 [230.0 to 18061.0] | 1906.95 [357.0 to 4200.0] | 2078.40 [487.0 to 13553.9] | 1983.90 [230.0 to 18061.0]
  Baseline (BL): number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Baseline (BL) | 1865.20 [459.0 to 5015.0] | 2202.22 [230.0 to 18061.0] | 1906.95 [357.0 to 4200.0] | 2078.40 [487.0 to 13553.9] | 1983.90 [230.0 to 18061.0]
  Change from BL Day7: number analyzed (Participants) | 14 | 29 | 8 | 9 | 60
  Change from BL Day7 | -146.50 [-721.4 to 710.0] | 377.80 [-1468.0 to 522220.0] | 22735.10 [-330.0 to 182380.0] | 23788.71 [-161.0 to 269529.0] | 358.90 [-1468.0 to 269529.0]
  Change from BL Day 14: number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Change from BL Day 14 | -321.30 [-2035.1 to 520.0] | 861.50 [-3483.3 to 59435.9] | 10728.40 [1262.0 to 104170.0] | 18580.01 [707.0 to 110421.6] | 973.00 [-3483.3 to 110421.6]
  Change from BL Day 21: number analyzed (Participants) | 14 | 29 | 8 | 8 | 59
  Change from BL Day 21 | 58.00 [-2302.0 to 524.0] | 331.00 [-3571.6 to 43336.0] | 3299.85 [-600.0 to 121100.0] | 3199.00 [-17.0 to 12957.4] | 490.00 [-3571.6 to 121100.0]
  Change from BL Day 28: number analyzed (Participants) | 14 | 27 | 8 | 9 | 58
  Change from BL Day 28 | 121.10 [-2952.0 to 1510.0] | 283.00 [-6443. to 9879.0] | 1104.00 [-890.0 to 331000.0] | 1211.00 [-606.0 to 12957.4] | 280.50 [-6443.7 to 33100.0]
  Change from BL Month 3: number analyzed (Participants) | 11 | 23 | 5 | 7 | 46
  Change from BL Month 3 | -124.90 [-2418.0 to 1985.5] | -358.00 [-5415.0 to 7050.0] | -487.60 [-1500.0 to 8140.0] | -377.00 [-1808.2 to 2641.6] | -330.00 [-5415.0 to 8140.0]

38. Secondary Outcome: Key Inflammatory Markers and Cytokine Parameters in Blood Within 1 Month by Maximum Cytokine Release Syndrome (CRS) Grade: INF-gamma
Description: INF-gamma at Pre-infusion, baseline, and change from baseline for Days 7, 14, 21, 28, Month 3
Time Frame: Pre-infusion, Baseline, Day 7, Day 14, Day 21, Day 28, Month 3
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Median (Full Range); unit: pg/mL
Arm/Group | NO CRS | Grade 1/2 | Grade 3 | Grade 4 | All Participants
Number analyzed (Participants) | 14 | 31 | 8 | 11 | 64
pg/mL
  Pre-infusion: number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Pre-infusion | 29.63 [1.0 to 283.0] | 23.39 [1.0 to 242.8] | 15.73 [6.4 to 31.5] | 5.79 [2.5 to 34.1] | 20.22 [1.0 to 283.0]
  Baseline (BL): number analyzed (Participants) | 14 | 31 | 8 | 9 | 63
  Baseline (BL) | 29.63 [1.0 to 283.0] | 22.51 [1.0 to 242.8] | 15.73 [6.4 to 31.5] | 4.77 [1.0 to 34.1] | 15.75 [1.0 to 283.0]
  Change from BL Day7: number analyzed (Participants) | 14 | 31 | 8 | 10 | 63
  Change from BL Day7 | 0.47 [-167.9 to 140.6] | 52.59 [-201.2 to 39452.4] | 3023.82 [-14.7 to 162376.0] | 1347.48 [60.2 to 89599.0] | 72.09 [-201.2 to 162376.0]
  Change from BL Day 14: number analyzed (Participants) | 13 | 30 | 8 | 9 | 60
  Change from BL Day 14 | -5.10 [-278.3 to 39.2] | -4.44 [-194.8 to 131.1] | 58.65 [-14.3 to 1328.7] | 102.04 [-2.2 to 8925.9] | 1.32 [-278.3 to 8925.9]
  Change from BL Day 21: number analyzed (Participants) | 13 | 29 | 8 | 8 | 58
  Change from BL Day 21 | -4.97 [-264.0 to 58.5] | 1.06 [-219.7 to 1384.6] | 0.53 [-22.8 to 1048.7] | 5.23 [-4.0 to 167.1] | -0.89 [-264.0 to 1384.6]
  Change from BL Day 28: number analyzed (Participants) | 14 | 28 | 8 | 9 | 59
  Change from BL Day 28 | -6.93 [-269.9 to 60.4] | 0.20 [-223.6 to 738.8] | -1.19 [-26.1 to 187.7] | 0.36 [-4.7 to 138.4] | -0.62 [-269.9 to 738.8]
  Change from BL Month 3: number analyzed (Participants) | 11 | 22 | 6 | 6 | 45
  Change from BL Month 3 | -6.08 [-278.6 to 167.5] | -14.58 [-173.9 to 7.6] | 21.25 [-7.7 to 37.2] | -0.67 [-4.4 to 23.1] | -5.71 [-278.6 to 167.5]

39. Secondary Outcome: Key Inflammatory Markers and Cytokine Parameters in Blood Within 1 Month by Maximum Cytokine Release Syndrome (CRS) Grade: Interleukin-6 (IL-6)
Description: IL-6 at Pre-infusion, baseline, and change from baseline for Days 7, 14, 21, 28, Month 3
Time Frame: Pre-infusion, Baseline, Day 7, Day 14, Day 21, Day 28, Month 3
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Median (Full Range); unit: pg/mL
Arm/Group | NO CRS | Grade 1/2 | Grade 3 | Grade 4 | All Participants
Number analyzed (Participants) | 14 | 31 | 8 | 11 | 64
pg/mL
  Pre-infusion: number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Pre-infusion | 2.42 [0.4 to 12.0] | 2.89 [0.2 to 19.6] | 1.00 [0.8 to 9.4] | 2.27 [0.4 to 6.2] | 2.27 [0.2 to 19.6]
  Baseline (BL): number analyzed (Participants) | 14 | 31 | 8 | 10 | 63
  Baseline (BL) | 2.42 [0.4 to 12.0] | 2.83 [0.2 to 19.6] | 1.00 [0.8 to 9.4] | 1.84 [0.2 to 6.2] | 1.99 [0.2 to 19.6]
  Change from BL Day7: number analyzed (Participants) | 14 | 31 | 8 | 10 | 63
  Change from BL Day7 | -0.23 [-9.6 to 4.3] | 2.64 [-13.1 to 61.3] | 52.75 [-0.6 to 7201.6] | 141.68 [1.3 to 12615.8] | 2.64 [-13.1 to 12615.8]
  Change from BL Day 14: number analyzed (Participants) | 13 | 30 | 8 | 9 | 60
  Change from BL Day 14 | -0.36 [-2.3 to 4.1] | -0.67 [-13.4 to 21.5] | 8.88 [-0.6 to 30.4] | 165.16 [-0.2 to 5734.8] | -0.11 [-13.4 to 5734.8]
  Change from BL Day 21: number analyzed (Participants) | 13 | 29 | 8 | 8 | 58
  Change from BL Day 21 | -0.97 [-5.3 to 5.3] | -0.46 [-15.4 to 103.4] | 1.65 [-0.6 to 265.2] | 50.75 [-0.2 to 5734.8] | -0.09 [-15.4 to 5734.8]
  Change from BL Day 28: number analyzed (Participants) | 14 | 28 | 8 | 9 | 59
  Change from BL Day 28 | -0.98 [-7.8 to 1.9] | -0.28 [-17.5 to 33.0] | 0.91 [-0.6 to 138.6] | 38.13 [-0.0 to 2148.4] | -0.03 [-17.5 to 2148.4]
  Change from BL Month 3: number analyzed (Participants) | 11 | 22 | 6 | 6 | 45
  Change from BL Month 3 | 0.34 [-10.8 to 22.7] | -0.59 [-8.9 to 1.2] | 0.56 [-0.6 to 30.3] | 0.40 [-0.9 to 3.2] | -0.19 [-10.8 to 30.3]

40. Secondary Outcome: Key Inflammatory Markers and Cytokine Parameters in Blood Within 1 Month by Maximum Cytokine Release Syndrome (CRS) Grade: Interleukin-2 (IL-2)
Description: IL-2 at Pre-infusion, baseline, and change from baseline for Days 7, 14, 21, 28, Month 3
Time Frame: Pre-infusion, Baseline, Day 7, Day 14, Day 21, Day 28, Month 3
Population: Safety set: All subjects who received an infusion of tisagenlecleucel
Measure: Median (Full Range); unit: pg/mL
Arm/Group | NO CRS | Grade 1/2 | Grade 3 | Grade 4 | All Participants
Number analyzed (Participants) | 14 | 31 | 8 | 11 | 64
pg/mL
  Pre-infusion: number analyzed (Participants) | 14 | 30 | 8 | 9 | 61
  Pre-infusion | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3]
  Baseline (BL): number analyzed (Participants) | 14 | 31 | 8 | 10 | 63
  Baseline (BL) | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.3]
  Change from BL Day7: number analyzed (Participants) | 14 | 31 | 8 | 10 | 63
  Change from BL Day7 | 3.33 [0.0 to 6.7] | 3.15 [0.0 to 7.0] | 13.14 [5.0 to 63.7] | 7.48 [2.9 to 12.1] | 5.16 [0.0 to 63.7]
  Change from BL Day 14: number analyzed (Participants) | 13 | 30 | 8 | 9 | 60
  Change from BL Day 14 | NA [NA to NA] — N/A = below limit of detection | 0.00 [0.00 to 0.00] | NA [NA to NA] — N/A = below limit of detection | 4.56 [4.56 to 4.6] | 0.00 [0.0 to 4.6]
  Change from BL Day 21: number analyzed (Participants) | 13 | 29 | 8 | 8 | 58
  Change from BL Day 21 | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection
  Change from BL Day 28: number analyzed (Participants) | 14 | 28 | 8 | 9 | 59
  Change from BL Day 28 | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection
  Change from BL Month 3: number analyzed (Participants) | 11 | 22 | 6 | 6 | 45
  Change from BL Month 3 | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection | NA [NA to NA] — N/A = below limit of detection

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: Adverse events were collected during the post-infusion period (starting at the day of first infusion until the end of the study), up to maximum duration of 60 months for each patient.
Description: AE description: Any sign or symptom that occurs during the post-infusion period (starting at the day of first infusion of CTL019 until the end of the study).
Arm/Group | Tisagenlecleucel (CTL019) - All Participants
All-Cause Mortality (participants affected / at risk) | 30/64
Serious Adverse Events (participants affected / at risk) | 52/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel (CTL019) - All Participants (N=64)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 23
Neutropenia (Blood and lymphatic system disorders) | 3
Atrioventricular block second degree (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Papilloedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Physical deconditioning (General disorders) | 1
Pyrexia (General disorders) | 7
Cytokine release syndrome (Immune system disorders) | 41
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1
Bacterial sepsis (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis of male external genital organ (Infections and infestations) | 1
Cholecystitis infective (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 3
Corona virus infection (Infections and infestations) | 1
Enterovirus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory syncytial virus infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Rotavirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic embolus (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Vascular device infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Transfusion related complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Embolic stroke (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 4
Headache (Nervous system disorders) | 1
Idiopathic intracranial hypertension (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel (CTL019) - All Participants (N=64)
Anaemia (Blood and lymphatic system disorders) | 27
Lymphopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Sinus tachycardia (Cardiac disorders) | 6
Tachycardia (Cardiac disorders) | 15
Periorbital oedema (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 27
Catheter site pain (General disorders) | 4
Chills (General disorders) | 10
Fatigue (General disorders) | 15
Pain (General disorders) | 4
Pyrexia (General disorders) | 21
Cytokine release syndrome (Immune system disorders) | 19
Hypogammaglobulinaemia (Immune system disorders) | 33
Gastroenteritis (Infections and infestations) | 4
Influenza (Infections and infestations) | 4
Otitis media (Infections and infestations) | 4
Rhinovirus infection (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 5
Activated partial thromboplastin time prolonged (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 21
Aspartate aminotransferase increased (Investigations) | 20
Blood bilirubin increased (Investigations) | 8
Blood creatinine increased (Investigations) | 9
Blood fibrinogen decreased (Investigations) | 4
Blood immunoglobulin M decreased (Investigations) | 4
International normalised ratio increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 16
Neutrophil count decreased (Investigations) | 28
Platelet count decreased (Investigations) | 20
Prothrombin time prolonged (Investigations) | 9
Weight decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 35
Decreased appetite (Metabolism and nutrition disorders) | 21
Hypernatraemia (Metabolism and nutrition disorders) | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 19
Hypophosphataemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 24
Anxiety (Psychiatric disorders) | 7
Confusional state (Psychiatric disorders) | 6
Acute kidney injury (Renal and urinary disorders) | 5
Haematuria (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 12
Hypotension (Vascular disorders) | 9

LIMITATIONS AND CAVEATS:
Safety data reported is based on all the 64 infused patients with data cutoff of 24May2019.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT02228096/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT02228096/SAP_001.pdf